CLINICAL TRIAL: NCT01146743
Title: Prospective Randomized Controlled Trial for Endoscopic Ultrasound Guided and Percutaneous Transhepatic Gallbladder Drainage for Acute Cholecystitis in High Risk Patients
Brief Title: Prospective Trial for Endoscopic Ultrasound Guided Gallbladder Drainage for Acute Cholecystitis in High Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: SangSooLee/professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUS_GB1
Record Dates: First submitted 2010-06-09; First posted 2010-06-22 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Cholecystitis
Keywords: EUS-guided transmural cholecystostomy
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EUS-guided (Active Comparator): EUS-guided gallbladder drainage in acute cholecystitis with high risk patients
  Interventions: Procedure: EUS-guided gallbladder drainage
- percutaneous transhepatic (Active Comparator): percutaneous transhepatic gallbladder drainage in acute cholecystitis with high risk patients
  Interventions: Procedure: percutaneous transhepatic gallbladder drainage

INTERVENTIONS:
Procedure: EUS-guided gallbladder drainage — EUS-guided gallbladder drainage was performed with a linear-array echoendoscope. The initial puncture was performed at the antrum of the stomach or bulb of the duodenum and was chosen to access the gallbladder body or neck and avoid visible vessels. After removal of the needle, a 6F or 7F bougie were inserted and then removed to dilate the tract. Afterward, nasobiliary drainage tube or stent was placed.
  Other Names: EUS-guided transmural drainage
  Arms: EUS-guided
Procedure: percutaneous transhepatic gallbladder drainage — Under ultrasound guidance, needle punctured to gallbladder via percutaneous transhepatic route.
  Other Names: percutaneous cholecystostomy
  Arms: percutaneous transhepatic

SUMMARY:
The investigators would like to conduct a prospective, randomized non-inferiority study to compare clinical outcome between endoscopic ultrasound (EUS) guided gallbladder drainage and percutaneous transhepatic gallbladder drainage (PTGBD) in high risk acute cholecystitis patients.

DETAILED DESCRIPTION:
The primary outcome is to compare clinical resolution rate of EUS-guided gallbladder drainage versus percutaneous transhepatic gallbladder drainage in acute cholecystitis patients with high risk.

The secondary outcome is to compare complications, conversion rate to open cholecystectomy during laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* high risk for general anesthesia and emergency operation (American Society of Anesthesiologists, ASA grade III or IV)

Exclusion Criteria:

* Age below 18 years
* Pregnancy
* When the risks of endoscopy to patient are judged to outweigh the most favorable benefits of the procedure.
* Unstable or unwilling to comply with follow-up
* When a perforated viscus is known or suspected
* Simultaneously participating in another investigational drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Clinical response rate | Within 72 hours from procedure
  Definition of clinical response rate within 72 hours from procedure was improvement of local signs and systemic signs of inflammation.

SECONDARY OUTCOMES:
Complication rate | Complications during the procedure or within 1 weeks
  Complication was defined as any procedure-related complications during the procedure or within 1 week, including bile leakage, pneumoperitoneum, bleeding, and etc.
Conversion rate | During laparoscopic cholectstectomy
  Conversion was defined as conversion to open cholecystectomy during laparoscopic cholecystectomy.

CONTACTS AND LOCATIONS:
Overall Officials: SangSoo Lee, M.D., Study Director — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Lee SS, Park DH, Hwang CY, Ahn CS, Lee TY, Seo DW, Lee SK, Kim MW. EUS-guided transmural cholecystostomy as rescue management for acute cholecystitis in elderly or high-risk patients: a prospective feasibility study. Gastrointest Endosc. 2007 Nov;66(5):1008-12. doi: 10.1016/j.gie.2007.03.1080. Epub 2007 Sep 4. PMID 17767933